CLINICAL TRIAL: NCT05500300
Title: Effects on Isometric Force Induction, Tolerance and Fatigue of Neuromuscular Electrical Stimulation and High Intensity Focused Electromagnetic Field in Healthy Subjects
Brief Title: Electrical Stimulation With Different Currents and Electromagnetic Fields
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maimonides University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 5891
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Healthy
Keywords: Electrical stimulation; Muscle Strength; Fatigue; Assessments, pain; Electromagnetic Fields; Physiotherapy
MeSH Terms: conditions — Fatigue; Pain

STUDY DESIGN:
Intervention Model Description: 30 male subjects will receive 4 types of electrical stimulation (Aussie, Neo-Russian, Rectangular biphasic symmetric waveform, Rectangular biphasic symmetric waveform with intra-pulse interval) and High Intensity Focused Electromagnetic Field (HIFEM) in a randomized order.
  Maximal voluntary isometric contraction (MVIC) and maximal elicited induced contraction (MEIC) will be measured with an isometric dynamometer. The best rep will be used. Whenever the third one is the best, additional measurements will be taken until a decrease in torque is obtained to determine the maximum. MVIC will be used for data normalization.
  The Visual Analogue Scale (VAS) will be used to assess tolerance to treatment. One week later, subjects will receive, randomly, a fatigue protocol with the 4 types of electrical stimulation and the HIFEM, which consists in 21 reps. A fatigue index (FI) will be calculated.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Neo-Russian Electrical Stimulation (Experimental): Subjects will receive Neo-Russian electrical stimulation. The Maximal Elicited Induced Contraction (MEIC) will be measured.
  One week later, after a washout period, a fatigue will be done with this type of current.
  Interventions: Device: Neo-Russian
- Aussie Electrical Stimulation (Experimental): Subjects will receive Aussie electrical stimulation. The Maximal Elicited Induced Contraction (MEIC) will be measured.
  One week later, after a washout period, a fatigue will be done with this type of current.
  Interventions: Device: Aussie
- RBS Electrical Stimulation (Experimental): Subjects will receive RBS electrical stimulation. The Maximal Elicited Induced Contraction (MEIC) will be measured.
  One week later, after a washout period, a fatigue will be done with this type of current.
  Interventions: Device: RBS
- RBS-IPI Electrical Stimulation (Experimental): Subjects will receive RBS-IPI electrical stimulation. The Maximal Elicited Induced Contraction (MEIC) will be measured.
  One week later, after a washout period, a fatigue will be done with this type of current.
  Interventions: Device: RBS-IPI
- HIFEM (Experimental): Subjects will receive HIFEM electrical stimulation. The Maximal Elicited Induced Contraction (MEIC) will be measured.
  One week later, after a washout period, a fatigue will be done with this type of current.
  Interventions: Device: HIFEM

INTERVENTIONS:
Device: Neo-Russian — Subjects will receive Neo-Russian electrical stimulation with three reps (5 sec work x 60 sec rest), and the Maximal Electrical Induced Contraction (MEIC) will be measured.
  They will be asked how uncomfortable the stimulation was, using Visual Analogue Scale (VAS).
  One week later, subjects will receive a fatigue protocol that consists in 21 reps (5 sec work x 5 sec rest), and the Maximal Electrical Induced Contraction (MEIC) will be measured for each contraction.
  Arms: Neo-Russian Electrical Stimulation
Device: Aussie — Subjects will receive Aussie electrical stimulation with three reps (5 sec work x 60 sec rest), and the Maximal Electrical Induced Contraction (MEIC) will be measured.
  They will be asked how uncomfortable the stimulation was, using Visual Analogue Scale (VAS).
  One week later, subjects will receive a fatigue protocol that consists in 21 reps (5 sec work x 5 sec rest), and the Maximal Electrical Induced Contraction (MEIC) will be measured for each contraction.
  Arms: Aussie Electrical Stimulation
Device: RBS — Subjects will receive RBS electrical stimulation with three reps (5 sec work x 60 sec rest), and the Maximal Electrical Induced Contraction (MEIC) will be measured.
  They will be asked how uncomfortable the stimulation was, using Visual Analogue Scale (VAS).
  One week later, subjects will receive a fatigue protocol that consists in 21 reps (5 sec work x 5 sec rest), and the Maximal Electrical Induced Contraction (MEIC) will be measured for each contraction.
  Arms: RBS Electrical Stimulation
Device: RBS-IPI — Subjects will receive RBS-IPI electrical stimulation with three reps (5 sec work x 60 sec rest), and the Maximal Electrical Induced Contraction (MEIC) will be measured.
  They will be asked how uncomfortable the stimulation was, using Visual Analogue Scale (VAS).
  One week later, subjects will receive a fatigue protocol that consists in 21 reps (5 sec work x 5 sec rest), and the Maximal Electrical Induced Contraction (MEIC) will be measured for each contraction.
  Arms: RBS-IPI Electrical Stimulation
Device: HIFEM — Subjects will receive HIFEM electrical stimulation with three reps (5 sec work x 60 sec rest), and the Maximal Electrical Induced Contraction (MEIC) will be measured.
  They will be asked how uncomfortable the stimulation was, using Visual Analogue Scale (VAS).
  One week later, subjects will receive a fatigue protocol that consists in 21 reps (5 sec work x 5 sec rest), and the Maximal Electrical Induced Contraction (MEIC) will be measured for each contraction.
  Arms: HIFEM

SUMMARY:
Muscle strength is the amount of force generated by muscle contraction. It could be measured with an isometric dynamometer. This is a validated tool that could be used to measure Maximal Voluntary Isometric Contraction (MVIC) and Maximal Electrical Induced Contraction (MEIC). It is claimed that higher MEIC values will result in more force gained.

If a current is more tolerated it will be easier to achieve better MEIC values. Tolerance to an electrical stimulation could be measured with the Visual Analogue Scale (VAS). A ratio between Normalized MEIC / VAS is often used, implying that the current is better with a higher ratio.

Muscle fatigue is defined as a temporary loss or decrease in force-generating ability due to previous contractions. It is claimed that medium frequency neuromuscular electrical stimulation (NMES) generates more fatigue than low frequency currents.

Aussie is a medium-frequency alternating current, sinusoidal waveform, 1 KHz carrier frequency.

Neo-Russian is a medium-frequency current, rectangular biphasic symmetrical waveform, 2,5 KHz carrier frequency.

Rectangular Biphasic symmetrical (RBS) waveform is a type of Low Pulsed Current (LPC), claimed to be better than classical Russian Current.

Purpose:

As it has been claimed that LPC is better in MEIC and tolerance, the aim of this study is to compare it with two newer medium frequency currents in terms of MEIC, tolerance and fatigue.

Methods:

Thirty male subjects, right leg dominant, will receive randomly the 3 types of electrical stimulation. Before that, the MVIC will be measured for data normalization.

The MVIC and MEIC will be measured with an isometric dynamometer. In both measurements, subjects will be asked to perform three reps (5 sec work x 120 sec rest) and the best one will be used. Whenever the third one was the best, additional measurements will be taken until a decrease in torque will be obtained to determine the maximum.

To apply Aussie electrical stimulation, an Aussie Sport (Ibramed) will be used. To apply Neo-Russian, a Neurodyn III (Ibramed) will be used. To apply RBS, a Genesy (Globus) will be used.

The VAS will be used to assess tolerance to each treatment. One week later, the subjects will receive, randomly, a fatigue protocol that consists in 21 reps (5 sec work x 5 sec rest) of electrical stimulation with the three types of current. The data will be normalized with the MVIC and the reps equal or below 50 % of the first rep will be considered as a fatigue rep.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Male
* Right leg dominant
* Exercising regularly

Exclusion Criteria:

* History of injuries in the right leg
* Skin lesions
* Having a pacemaker
* Having a cardiovascular disease.
* Having a neurological disorder.
* Exercise 72 h before the procedure.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-22 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Maximal Voluntary Isometric Contraction (MVIC) | Day 1
  Force generated by the patient during a maximal voluntary isometric contraction, measured by an isometric dynamometer with load cell and computer interface.
  The best of the 3 repetitions will be considered. Whenever the third one is the best, additional measurements will be taken until a decrease in torque is obtained in order to determine the maximum.
  Unit: Newtons (N)
Maximal Electrical Induced Contraction (MEIC) | Day 1
  Force generated in the muscle while applying electrical stimulation and HIFEM, measured by an isometric dynamometer with load cell and computer interface. This data (in Newtons) will be normalized with the MVIC.
  Unit: percentage of MVIC
Visual Analogue Scale | Day 1
  Visual Analogue Scale (VAS): Magnitude of pain, marked in a analogue scale by participants, to determine how unpleasant is each type of stimulation (applied in randomized order).
  Expresed in centimeters.
  * Minimum value: 0
  * Maximum value: 10
  * A higher score implicates a worse outcome. VAS wil be evaluated 5 times, 1 per type of stimulation.

SECONDARY OUTCOMES:
Fatigue index | Day 7
  The MEIC decrease between the first and the 21st rep, previously normalized with the MVIC.
  * Minimum value: -1
  * Maximum value: 1
  * The lower the value, the greater the fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Maimonides University, Buenos Aires, Buenos Aires F.D., Argentina